CLINICAL TRIAL: NCT01684163
Title: Phase 2, Double-Blind, Placebo Controlled, Randomized Withdrawal, Parallel Efficacy and Safety Study of GLYX-13 in Subjects With Inadequate/Partial Response to Antidepressants During the Current Episode of Major Depressive Disorder
Brief Title: Efficacy and Safety of GLYX-13 in Subjects With Inadequate/Partial Response to Antidepressants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLYX13-C-202
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Major Depressive Disorder
Keywords: depression; MDD; GLYX-13; HDRS-17; HAMD-17
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo injection (Placebo Comparator): Normal saline
  Interventions: Drug: Placebo
- GLYX-13, 5 mg/kg (Experimental): Low dose of GLYX-13
  Interventions: Drug: GLYX-13 5 mg/kg
- GLYX-13, 10 mg/kg (Experimental): High dose of GLYX-13
  Interventions: Drug: GLYX-13 10 mg/kg

INTERVENTIONS:
Drug: GLYX-13 5 mg/kg — Intravenous administration of 5 mg/kg into arm.
  Other Names: GLYX-13 IV Dose
  Arms: GLYX-13, 5 mg/kg
Drug: GLYX-13 10 mg/kg — Intravenous administration of 10 mg/kg into arm.
  Other Names: GLYX-13 IV Dose
  Arms: GLYX-13, 10 mg/kg
Drug: Placebo — Intravenous administration of normal saline into arm.
  Other Names: Normal Saline
  Arms: Placebo injection

SUMMARY:
GLYX-13 is a NMDA receptor glycine site partial agonist being studied in subjects with major depressive disorder (depression) who have responded inadequately to another antidepressant drug during the current episode. This trial will assess the effects of GLYX-13 on depression when added to another antidepressant drug that the patient is already taking.

DETAILED DESCRIPTION:
To evaluate the mean difference in Hamilton Depression Rating Scale 17 (HDRS-17) score for the combined GLYX-13 mean change versus the placebo group mean change at the end of a 6 week randomized withdrawal phase (predose baseline score - score at end of randomized withdrawal period).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Aged 18 to 65 years
* Meets DSM-IV-TR) criteria for major depressive disorder (MDD)
* Current episode has lasted ≥ 8 weeks before Screening with an inadequate response to all approved antidepressant agent(s) administered at an adequate dose and duration for the current episode
* Taking no antidepressant agent currently or taking an SSRI or SNRI
* HDRS-17 score ≥ 18 at screening and predose baseline
* Female subjects of childbearing potential with a negative serum pregnancy test prior to entry into the study and who are practicing an adequate method of birth control and who do not plan to become pregnant during the course of the study.
* Clinical laboratory values < 2 times the upper limit of normal (ULN) or deemed not clinically significant per the investigator and Naurex medical monitor
* Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments
* Based on the investigator and Naurex medical monitor's clinical judgment, subjects with eating disorders, obsessive compulsive disorder (OCD), panic disorder, post-traumatic stress disorder (PTSD), and generalized anxiety disorders secondary to major depressive episodes (MDEs) are permitted.

Exclusion Criteria:

* Axis I diagnosis of delirium, dementia, dysthymia, amnestic or other cognitive disorder, schizophrenia or other psychotic disorder, bipolar I or II disorder, eating disorder (anorexia or bulimia nervosa), obsessive-compulsive disorder, panic disorder, acute stress disorder, agoraphobia, social phobia, attention-deficit hyperactivity disorder (ADHD), or PTSD
* A clinically significant current Axis II diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder
* Experiencing hallucinations, delusions, or any psychotic symptomatology in the current episode; lifetime history of psychosis
* Huntington's, Parkinson's, Alzheimer's, Multiple Sclerosis, or a history of seizures or strokes
* Currently hospitalized or residing in an in-patient facility during the study participation
* Substance abuse within the last 12 months
* Women who are planning to become pregnant during the course of the study
* Allergy or intolerance to current antidepressant or other current medications
* Participation in any clinical trial of an investigational product or device within 30 days of enrollment in this trial with the exception of GLYX13-C-201.
* Positive screen for drugs of abuse
* Have received electroconvulsive therapy, transcranial magnetic stimulation (TMS), or vagal nerve stimulation (VNS) for the current depressive episode
* Pose current (past 6 months) suicide risk based on administration of the C SSRS and the investigator's clinical judgment
* Human immunodeficiency virus (HIV) infection (based on the HIV-1 & HIV-2 antibody screen) or other ongoing infectious disease
* Females who are currently pregnant or planning to become pregnant during the course of the study
* Dextromethorphan or tramadol since these are serotonin uptake inhibitors
* History of allergy, sensitivity, or intolerance to N-methyl-D-aspartate receptor [NMDAR] ligands

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale Score | 6 weeks, 12 weeks, 16 weeks

SECONDARY OUTCOMES:
Clinical Global Impression of Change | 6 weeks, 12 weeks, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Naurex Inc, an affilate of Allergan plc
Locations (26):
- United States (26):
  - University of Alabama Office of Psychiatric Clinical Research, Birmingham, Alabama
  - Pharmacology Research Institute, Encino, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pacific Institute of Medical Research, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Evanston Premier Healthcare Research, LLC, Northbrook, Illinois
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - University of Kansas, Wichita, Kansas
  - PharmaSite Research , Inc., Baltimore, Maryland
  - Bostin Clinical Trials, Inc., Roslindale, Massachusetts
  - CRI Lifetree, Marlton, New Jersey
  - Global Medical Institutes LLC, Princeton, New Jersey
  - Clinilabs, Inc., New York, New York
  - Michael R Liebowitz MD, New York, New York
  - Finger Lake Clinical Research, Rochester, New York
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - CRI Lifetree, Phildadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center of Dallas, Dallas, Texas
  - CRI Lifetree, Salt Lake City, Utah
  - Summit Research Network, Seattle, Washington